CLINICAL TRIAL: NCT03267797
Title: Intrauterine Administration of Autologous hCG-activated Peripheral Blood Mononuclear Cells Improves Pregnancy Outcomes in Patients With Recurrent Implantation Failure; a Double-blind Randomized Control Trial Study
Brief Title: hCG-activated PBMC-therapy in RIF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SCARM Institute, Tabriz, Iran (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCARM-infertility-004
Record Dates: First submitted 2017-08-27; First posted 2017-08-30 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Recurrent Implantation Failure
Keywords: Recurrent Implantation Failure; Peripheral blood mononuclear cell; Human chorionic gonadotropin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and the person who analyzed the results were blinded in this study. Participants were aware of the study before being randomized and informed consent was obtained from them. It should be noted that the person analyzing the results had no other role in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Peripheral blood mononuclear cells (PBMCs) were administered into the uterine cavity of RIF patients in this group.
  Interventions: Other: Peripheral Blood Monouclear Cell
- Control group (Placebo Comparator): Phosphate buffer saline (PBS) as placebo was injected into the uterine cavity of RIF patients in this group.
  Interventions: Other: Phosphate Baffer Saline

INTERVENTIONS:
Other: Peripheral Blood Monouclear Cell — Blood samples (20 mL) were taken from individual patients at the time of ovulation induction. Then PBMC were isolated and cultured (20-30 million cells) 48 hour at the presence of hCG (10IU/ml daily). Afterward,15-20 million PBMCs in 500 microlitres PBS were injected into the uterine cavity two days before embryo transfer (ET) using ET catheter.
  Other Names: PBMC
  Arms: Treatment group
Other: Phosphate Baffer Saline — Only 500 microlitres PBS will be injected into the uterine cavity, instead of PBMCs, two days before embryo transfer (ET) using ET catheter.
  Other Names: PBS
  Arms: Control group

SUMMARY:
Despite the many research done in the field of infertility and in vitro fertilization (IVF), more than half of the embryos transmitted in the IVF and intracytoplasmic sperm injection (ICSI) do not implant successfully. Currently, pregnancy failure following at least three IVF/ET cycle, so that one or two high-quality embryos transmitted in each cycle is defined as recurrent implantation failure (RIF). Maternal and fetal factors can be a reason for implantation failure; maternal factors include endometrial receptivity, uterine anatomic abnormalities, and immunologic factors. Implantation failure with embryonic reasons includes genetic abnormalities and any factor that affects the implantation and growth of the embryo within the uterus. In recent years, the involvement of immune-related factors mainly natural killer cells (NK), dendritic cells (DCs), macrophages (MQ), regulatory T cells (Treg) and Th-1, in the endometrial differentiation and development and endometrial receptivity, as well as induction of immunological tolerance to the fetus, have been reported.

DETAILED DESCRIPTION:
248 women with the history of implantation failure volunteered to receive PBMC-therapy. After immunologic consultation and doing flow cytometry analysis, 100 women with at least three IVF/ET failure who had low Th-17/Treg ratio in comparison with healthy control were enrolled in this study. These 100 patients divided randomly into two groups, 50 patients received PBMC and 50 patients as the control group received PBS. PBMCs were obtained from patients themselves five days before embryo transfer (ET) and were cultured with hCG for 48 hours. Frothy-eight hours later, PBMCs were then administered into the uterine cavity of that patient from the study group two days before ET. PBS was inseminated into the uterine cavity of the control group instead of PBMC. The concentration of inflammatory cytokines was examined in the supernatant of cultured PBMCs 2, 24 and 48 hour after incubation by ELISA. The pregnancy occurrence was confirmed 12 days after ET through positive pregnancy test (β-hCG test). The success of implantation and the occurrence of clinical pregnancy were evaluated by ultrasound through the observation of the number and the location of gestational sacs at 5-6 weeks and confirming the embryo heart pulsation.

ELIGIBILITY:
All patients were evaluated in accordance with the following inclusion and exclusion criteria;

Inclusion Criteria:

1. Having at least three implantation failures following IVF
2. Having primary infertility
3. Age under 45 years old
4. Having regular menstrual cycles
5. BMI under 30

Exclusion Criteria:

1. Having polycystic ovary syndrome
2. The presence of uterine pathology;
3. Poor ovarian reserve
4. Having chromosomal abnormalities
5. Presence of auto anti-bodies such as anti-TPO, anti-TG, ACA, APA, ANA, and anti-dsDNA
6. Presence of mutations involving the coagulation system such as deficiency of factor XII, Pro C, Pro S
7. Positive HIV, HCV or HBV tests

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-07 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
pregnancy occurrence | "12 days after embryo transfer"
  Laboratory tests (beta-hCG test)
examination of inflammatory cytokines (IL-1B, TNF-a and INF-Y) secretion levels in supernatant | "48 hours after culturing"
  ELISA technique

SECONDARY OUTCOMES:
Clinical pregnancy rate in patients with recurrent implantation failure (RIF) | "in 5-6 weeks"
  detection the number and location of gestational sacs by ultrasound
The live birth rate by patients with recurrent implantation failure (RIF) | "After about 9 months of positive βHCG test"
  By gynecologists and obstetricians will monitor
The miscarriage rate in patients with recurrent implantation failure (RIF) | "When ever during the pregnancy period (up to 9 months)"
  By gynecologists and obstetricians will monitor

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Nouri, Ph.D, Study Chair — Head of SCARM institute; Mehdi Yousefi, Ph.D, Study Director — SCARM institute
Locations (1):
- Valiasr Hospital, Tabriz, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chaouat G, Ledee-Bataille N, Zourbas S, Ostojic S, Dubanchet S, Martal J, Frydman R. Cytokines, implantation and early abortion: re-examining the Th1/Th2 paradigm leads to question the single pathway, single therapy concept. Am J Reprod Immunol. 2003 Sep;50(3):177-86. doi: 10.1034/j.1600-0897.2003.00080.x. PMID 14629021
- [Result] Simon A, Laufer N. Repeated implantation failure: clinical approach. Fertil Steril. 2012 May;97(5):1039-43. doi: 10.1016/j.fertnstert.2012.03.010. Epub 2012 Mar 30. PMID 22464086
- [Result] Hoozemans DA, Schats R, Lambalk CB, Homburg R, Hompes PG. Human embryo implantation: current knowledge and clinical implications in assisted reproductive technology. Reprod Biomed Online. 2004 Dec;9(6):692-715. doi: 10.1016/s1472-6483(10)61781-6. PMID 15670421
- [Result] Tomassetti C, Meuleman C, Pexsters A, Mihalyi A, Kyama C, Simsa P, D'Hooghe TM. Endometriosis, recurrent miscarriage and implantation failure: is there an immunological link? Reprod Biomed Online. 2006 Jul;13(1):58-64. doi: 10.1016/s1472-6483(10)62016-0. PMID 16820110
- [Result] Bulmer JN, Longfellow M, Ritson A. Leukocytes and resident blood cells in endometrium. Ann N Y Acad Sci. 1991;622:57-68. doi: 10.1111/j.1749-6632.1991.tb37850.x. No abstract available. PMID 2064208
- [Result] Mosmann TR, Cherwinski H, Bond MW, Giedlin MA, Coffman RL. Two types of murine helper T cell clone. I. Definition according to profiles of lymphokine activities and secreted proteins. J Immunol. 1986 Apr 1;136(7):2348-57. PMID 2419430
- [Result] Chou CH, Chen SU, Shun CT, Tsao PN, Yang YS, Yang JH. Divergent endometrial inflammatory cytokine expression at peri-implantation period and after the stimulation by copper intrauterine device. Sci Rep. 2015 Oct 15;5:15157. doi: 10.1038/srep15157. PMID 26469146
- [Result] Kosaka K, Fujiwara H, Tatsumi K, Yoshioka S, Higuchi T, Sato Y, Nakayama T, Fujii S. Human peripheral blood mononuclear cells enhance cell-cell interaction between human endometrial epithelial cells and BeWo-cell spheroids. Hum Reprod. 2003 Jan;18(1):19-25. doi: 10.1093/humrep/deg002. PMID 12525435
- [Result] Ideta A, Sakai S, Nakamura Y, Urakawa M, Hayama K, Tsuchiya K, Fujiwara H, Aoyagi Y. Administration of peripheral blood mononuclear cells into the uterine horn to improve pregnancy rate following bovine embryo transfer. Anim Reprod Sci. 2010 Jan;117(1-2):18-23. doi: 10.1016/j.anireprosci.2009.04.004. Epub 2009 May 3. PMID 19467808
- [Result] Yu N, Yang J, Guo Y, Fang J, Yin T, Luo J, Li X, Li W, Zhao Q, Zou Y, Xu W. Intrauterine administration of peripheral blood mononuclear cells (PBMCs) improves endometrial receptivity in mice with embryonic implantation dysfunction. Am J Reprod Immunol. 2014 Jan;71(1):24-33. doi: 10.1111/aji.12150. Epub 2013 Aug 1. PMID 23909917
- [Result] Okitsu O, Kiyokawa M, Oda T, Miyake K, Sato Y, Fujiwara H. Intrauterine administration of autologous peripheral blood mononuclear cells increases clinical pregnancy rates in frozen/thawed embryo transfer cycles of patients with repeated implantation failure. J Reprod Immunol. 2011 Dec;92(1-2):82-7. doi: 10.1016/j.jri.2011.07.001. Epub 2011 Oct 27. PMID 22035703
- [Result] Nakayama T, Fujiwara H, Maeda M, Inoue T, Yoshioka S, Mori T, Fujii S. Human peripheral blood mononuclear cells (PBMC) in early pregnancy promote embryo invasion in vitro: HCG enhances the effects of PBMC. Hum Reprod. 2002 Jan;17(1):207-12. doi: 10.1093/humrep/17.1.207. PMID 11756389
- [Result] Yoshioka S, Fujiwara H, Nakayama T, Kosaka K, Mori T, Fujii S. Intrauterine administration of autologous peripheral blood mononuclear cells promotes implantation rates in patients with repeated failure of IVF-embryo transfer. Hum Reprod. 2006 Dec;21(12):3290-4. doi: 10.1093/humrep/del312. Epub 2006 Oct 4. PMID 17021188
- [Result] Al-Azemi M, Raghupathy R, Azizieh F. Pro-inflammatory and anti-inflammatory cytokine profiles in fetal growth restriction. Clin Exp Obstet Gynecol. 2017;44(1):98-103. PMID 29714875
- [Result] Granot I, Gnainsky Y, Dekel N. Endometrial inflammation and effect on implantation improvement and pregnancy outcome. Reproduction. 2012 Dec;144(6):661-8. doi: 10.1530/REP-12-0217. Epub 2012 Oct 1. PMID 23028125